CLINICAL TRIAL: NCT05837273
Title: The Feasibility Usability and Effectiveness of Fully Immersive Horticultural-based Virtual Reality Cognitive Training for Community-dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202300244B0
Record Dates: First submitted 2023-03-28; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-03

CONDITIONS: Fully Immersive Virtual Reality
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fully immersive leisure-based virtual reality (Experimental)
  Interventions: Device: Fully-immersive VR
- Conventional cognitive training (Experimental)
  Interventions: Behavioral: Cognitive training
- control group (No Intervention)

INTERVENTIONS:
Device: Fully-immersive VR — For fully-immersive VR sets the highest level of immersion of VR technologies, presenting improvement in cognitive function in cognitive decline seniors. Fully immersive VR-based cognitive training also has a positive effect on psychological performance.
  Arms: Fully immersive leisure-based virtual reality
Behavioral: Cognitive training — For the cognitive training, the therapy is a non-pharmacological approach, used for a series of standardized tasks to maintain or even increase person's cognitive function. The therapy can effectively improve multiple cognitive performance, such as: attention, reaction time (processing speed), working memory, and visual-spatial ability.
  Arms: Conventional cognitive training

SUMMARY:
The pilot study will be a novel investigation of the usability and feasibility of leisure activities-based fully immersive VR cognitive training systems for cognitive training. We will recruit healthy aged individuals and occupational therapists for usability plus feasibility evaluation and perform the comparison of the effect with the developed VR intervention on psychological, daily life function and quality of life outcomes in populations experiencing cognitive decline. The fully-immersive VR system applied with horticultural therapy will be conducted in cognitive training and it was equipped with a headset and a pair of controllers for motion estimation and monitoring in a virtual environment. The findings of the research will effectively lead to advancement of the fully immersive leisure-based virtual reality cognitive training for elderly with cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Occupational therapists

  1. Have clinical experience for more than one year
* Healthy aged Individuals:

  1. An initial MoCA scores ≧ 20
  2. age between 60 to 85
  3. ability to follow instructions and perform tasks
  4. willing to provide written informed consent

Exclusion Criteria:

* Occupational therapists

  1. History of severe dizziness or epilepsy
  2. Unstable physical conditions accompanied by neurological or other orthopedic diseases may affect immersive VR experience
  3. Recent diagnosis of psychiatric disorders
* Healthy aged individuals:

  1. An initial MoCA scores lower than 20
  2. History of psychiatric disorders, major perceptual (visual or auditory) impairments, migraine or epilepsy, motion-sickness sensitive, unable to provide informed written consent due to severe cognitive impairment

[Effect study]

Inclusion Criteria:

1. An initial MoCA scores ≧ 20
2. age between 60 to 85
3. ability to follow instructions and perform tasks
4. willing to provide written informed consent

Exclusion Criteria:

1. An initial MoCA scores lower than 20
2. History of psychiatric disorders, major perceptual (visual or auditory) impairments, migraine or epilepsy, motion-sickness sensitive, unable to provide informed written consent due to severe cognitive impairment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment | baseline, after the intervention eight weeks, and at 3-month follow-up
  The Montreal Cognitive Assessment (MoCA) will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Wechsler Memory Scale | baseline, after the intervention eight weeks, and at 3-month follow-up
  Including Faces Recognition (total scale=48), Verbal Paired Associates (total scale = 32), Word Lists (total scale = 48), and Spatial Span (total scale=32) will be used to assess the immediate, delayed, and working memory tests. For each subtest, a higher number indicates better performance in memory function. The raw score of subtests will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Color trials test | baseline, after the intervention eight weeks, and at 3-month follow-up
  For Part 1, the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2, the respondent rapidly connects numbered circles in sequence, but alternates between pink and yellow. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors.
Change scores of Stroop test | baseline, after the intervention eight weeks, and at 3-month follow-up
  The participants will be tested under congruent and incongruent conditions. In the congruent condition, the participant will name the color ink of a word which is consistent with the written color name; whereas in the incongruent condition the participant will name the color ink differs from the written color name. The time to complete the task will be calculated for each condition

SECONDARY OUTCOMES:
Change scores of Wechsler Adult Intelligence Scale; WAIS | baseline, after the intervention eight weeks, and at 3-month follow-up
  The digit symbol test involves a key consisting of the numbers 1-9, each paired with a unique, easy-to-draw symbol such as a "V", "+" or ">".
  Matrix Reasoning
  This is a nonverbal reasoning task in which individuals are asked to identify patterns in designs. This subtest measures:
  non-verbal reasoning skills broad visual intelligence perceptual organization skills
Change scores of the short (12-item) form of the Everyday Cognition Scale (ECog-12) | baseline, after the intervention eight weeks, and at 3-month follow-up
  The short (12-item) form of the Everyday Cognition Scale (ECog-12), which was developed as an informant-rated report of cognitively mediated functional abilities in older adults. The ECog-12 asks participants to rate their current ability to perform cognitively mediated daily tasks related to everyday memory, language, visuospatial abilities, and executive functions compared with their ability to do the same task 10 years ago. Items are rated on a scale of 1-4, with 1 = Better or no change and 4 = Consistently much worse. The global, executive, and memory ECog-12 sub-domain scores were generated by averaging over the component items (sum of items/number of items) to maintain a range of 1 to 4 (with higher scores reflecting greater self-reported SCD).
Change scores of Amsterdam Instrumental Activity of Daily Living,A-IADL | baseline, after the intervention eight weeks, and at 3-month follow-up
  The Amsterdam Instrumental Activity of Daily Living (A-IADL) is an adaptive and computerized questionnaire designed to assess impairments in instrumental activities of daily living (IADL) in (early) dementia. The questionnaire is completed by a caregiver, such as a relative or friend.
  Each item has a 5-point scale response option (scored 0-4). The scoring of the Amsterdam Instrumental Activity of Daily Living is calculated using item response theory .Lower scores indicating poorer performance.
Change scores of the World Health Organization Quality of Life-Old(WHOQOL-OLD | baseline, after the intervention eight weeks, and at 3-month follow-up
  The World Health Organization Quality of Life-Old questionnaires demonstrate acceptable psychometric performance in a convenience sample of Taiwan older people. It are valuable measures of Quality of Life-Old for use with older people.Time frame for assessment is the past two weeks.
  The items are distributed into 4 domains (physical; psychological, social and environmental health) and 25 facets.
Change scores of WHOQOL-bref Taiwan Version | baseline, after the intervention eight weeks, and at 3-month follow-up
  As with the standard WHOQOL-BREF questionnaires the WHOQOL-BREF Taiwan version was simplified from the WHOQOL long form for Taiwan. For the purpose of cross-cultural comparison, the first 26 items were the same as the standard WHOQOL-BREF, which was developed from global studies. In addition to the 26 items, we applied the psychometric criteria proposed by the WHOQOL Group to select two more items from each of the two new facets to form the WHOQOL-BREF Taiwan version using data from the same 1,068 subjects. The selection process used for national items is described in the Results section. Thus, the WHOQOL-BREF Taiwan version contains 28 items classified into the same four domains as the standard WHOQOL-BREF. The scale administration and scoring procedures are the same as for the WHOQOL long form except that the facet score is based on only one item.
Change scores of Community Integration Questionnaire, CIQ | baseline, after the intervention eight weeks, and at 3-month follow-up
  The community integration questionnaire (CIQ) was designed to assess home integration, social integration and productive activity in persons with acquired brain injury. The instrument consists of 15 items and can be completed by self report or with the assistance of a family member or caregiver familiar with the person's health status and social activities.
Change scores of Geriatric Depression Scale (GDS) | baseline, after the intervention eight weeks, and at 3-month follow-up
  The Geriatric Depression Scale (GDS) - 15 items version is a self-administered questionnaire used to evaluate mood and depressive symptoms. The scores range is 0-15 and a score of 5 or greater taken as a possible indicator of depression.
Change scores of The Chinese Aging Well Profile (CAWP) | baseline, after the intervention eight weeks, and at 3-month follow-up
  It comprised eight open-ended questions focusing on the meaning and interpretation of 'subjective well-being', e.g., 'Can you tell me what the important contributors to your well-being are?', 'Can you describe the important elements in your life that make you feel happy?', 'Can you describe the important elements in your life that you dislike?' and 'What does well-being personally mean to you?' To adapt the Aging Well Profile for a Chinese population in Taiwan was secured. It was agreed that the new version would be called the Chinese Aging Well Profile (CAWP).
Change scores of Timed up and go (TUG) | baseline, after the intervention eight weeks, and at 3-month follow-up
  The TUG assesses the dynamic balance ability and mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers in frail elderly . The test-retest reliability of TUG on individuals with cognitive impairment was excellent .
Change scores of 30 second chair stand test,CST | baseline, after the intervention eight weeks, and at 3-month follow-up
  The 30 second sit-to-stand will be assessed to indicate the strength and endurance level of the lower extremities. The 30 second sit-to-stand was standardized to allow hand support during the rise to and descent from standing but required participants to let go of the armrests with each stand. The participants will be asked to stand up from a standardized chair and then sit down as many times as possible within 30 seconds. The feasibility and reliability of using sit-to-stand test in people with cognitive impairment have been established to be good.
Change scores of short physical performance battery,SPPB | baseline, after the intervention eight weeks, and at 3-month follow-up
  The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons. The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests . It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance). The SPPB has been shown to have predictive validity showing a gradient of risk for mortality, nursing home admission, and disability.
Change scores of International Physical Activity Questionnaires (IPAQ) | baseline, after the intervention eight weeks, and at 3-month follow-up
  The Chinese version of the International Physical Activity Questionnaires (IPAQ) is an international measure for health-related physical activity. A short form of IPAQ will be used to assess changes in physical activity before and after intervention in this study. The reliability and validity of IPAQ has been established across 12 countries .
  The self-report, short-form IPAQ , consists of three questions about days and time of vigorous, moderate, and walking activity in bouts of 10 min, with one question about daily sedentary time in the preceding seven days. The questionnaire was preceded by completion instructions and three questions about the types of vigorous, moderate, and light activity undertaken .
Change scores of The Clinical Frailty Scale (CFS) | baseline, after the intervention eight weeks, and at 3-month follow-up
  The aim of this scoping review is to identify and document the nature and extent of research evidence related to the Clinical Frailty Scale (CFS). The association of Clinical Frailty Scale (CFS) score with clinical outcomes highlights its utility in the care of the aging population.
  The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Change scores of Reported Edmonton Frail Scale (REFS) | baseline, after the intervention eight weeks, and at 3-month follow-up
  Reported Edmonton Frail Scale is an adaptation of Edmonton Frail Scale, that can be performed in less than 10 min by any healthcare professional. Reported Edmonton Frail Scale substitutes the last domain on Edmonton Frail Scale, the physical performance measure, with three self-assessed physical performance questions . This is ideal for use in busy cardiology clinics when patients are being assessed for suitability for intervention.Scoring for the Reported Edmonton Frail Scale range is 0 to18. Not Frail：0-5 ;Apparently Vulnerable：6-7; Mildly Frail：8-9;Moderate Frailty：10-11;Sever Frailty：12-18.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Taiwan